CLINICAL TRIAL: NCT02594254
Title: A Phase 2, Double-Blind, Placebo-Controlled and Open-Label Multi-Center Study to Evaluate the Microbiology and Safety of C16G2 Administered in Multiple Oral Gel Doses to Adult and Adolescent Dental Subjects
Brief Title: Phase 2 Study to Evaluate the Microbiology and Safety of C16G2 Administered to Adult and Adolescent Dental Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Collaborators: Vantage Data Designs, Inc. (Industry); SynteractHCR (Industry); Agility Clinical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3J15-203-00
Record Dates: First submitted 2015-10-28; First posted 2015-11-03 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Antimicrobial Peptides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Study Arm 1 (Experimental): Subjects in Study Arm 1 will receive 4 ml of 800 µM study drug administrations for a total of 28 consecutive days. Subjects will receive 4 C16G2 Gel or placebo administrations at the clinic on the first day, followed by morning (AM) and evening (PM) study drug administrations at the subjects' home for 27 consecutive days. Study drug will be administered via a manual brush.
  Interventions: Drug: C16G2 Gel; Other: Placebo
- Study Arm 2 (Experimental): Subjects in Study Arm 2 will receive 4 ml of 800 µM study drug administrations for a total of 28 consecutive days. Subjects will receive 4 C16G2 Gel or placebo administrations at the clinic on the first day, followed by morning (AM) and evening (PM) study drug administrations at the subjects' home for 27 consecutive days. Study drug will be administered via a manual brush and custom dental trays.
  Interventions: Drug: C16G2 Gel; Other: Placebo
- Study Arm 3 (Experimental): Subjects in open-label Study Arm 3 will receive 4 ml of 1600 µM study drug administrations for a total of 7 consecutive days. Subjects will receive 4 C16G2 Gel administrations at the clinic on the first day, followed by morning (AM) and evening (PM) study drug administrations at the clinic for 6 consecutive days. Study drug will be administered via a manual brush and custom dental trays.
  Interventions: Drug: C16G2 Gel
- Study Arm 4 (Experimental): Subjects in open-label Study Arm 4 will receive 4 ml 800 µM C16G2 Gel on a single day. Subjects will receive 4 study drug administrations at the clinic. Study drug will be administered via manual toothbrush and custom dental trays.
  Interventions: Drug: C16G2 Gel
- Study Arm 5 (Experimental): Subjects in open-label Study Arm 4 will receive 4 ml of 1600 µM C16G2 Gel on a single day. Subjects will receive 4 study drug administrations at the clinic. Study drug will be administered via manual toothbrush and custom dental trays.
  Interventions: Drug: C16G2 Gel
- Study Arm 6 (Experimental): If initiated, subjects in Study Arm 6 will receive 4 ml of 1600 µM study drug over a 7 day study drug administration period. Subjects will receive 4 C16G2 Gel or placebo administrations on the first day of dosing followed by morning (AM) and evening (PM) dosing for 6 consecutive days. Study drug will be administered via manual toothbrush and custom dental trays.
  Interventions: Drug: C16G2 Gel; Other: Placebo
- Study Arm 7 (Experimental): If initiated, subjects in Study Arm 7 will receive 4 ml of 800 µM or 1600 µM study drug on a single day once a week or once a month for a total of 4 days of C16G2 Gel or placebo administration. Subjects will receive 4 study drug administrations on the day of dosing. Study drug will be administered via manual toothbrush and custom dental trays.
  Interventions: Drug: C16G2 Gel; Other: Placebo

INTERVENTIONS:
Drug: C16G2 Gel — Antimicrobial peptide
  Other Names: Antimicrobial peptide
Other: Placebo — Placebo
  Arms: Study Arm 1; Study Arm 2; Study Arm 6; Study Arm 7

SUMMARY:
The purpose of this study is to evaluate if C16G2 Gel administered over a certain period of time either with a toothbrush or a custom dental tray can effectively kill bacteria in the mouth that cause dental cavities.

DETAILED DESCRIPTION:
This multi-center, multiple-arm study will evaluate the microbiological activity and safety of C16G2 Gel in male and female dental subjects, 12 to 75 years of age. The study will be conducted in a randomized, double-blind, placebo-controlled and open-label manner and enroll adolescent (12-17 years of age) and adult subjects (18-75 years of age).

A total of approximately 128 study subjects will be enrolled into up to 7 study arms. Study drug (C16G2 Gel or Placebo) will be administered via manual brush gel application (MBGA) or tray gel application (TGA). Two C16G2 concentrations will be evaluated. Four study arms will be conducted in a double blind manner, with a treatment allocation ratio of 4:1 (C16G2:Placebo), three study arms will be conducted in an open-label manner. Before dosing, eligible subjects will undergo professional dental prophylaxis on Day 0. Clinic visits for all study arms will include Visit 1 (Screening/Days -21 to 0), and a varying number of dosing and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 12-75 years of age, inclusive, at the time the Assent and/or Informed Consent Form is signed
2. Female subjects of childbearing potential, defined as not surgically sterile or at least two (2) years postmenopausal, must agree to use one of the following forms of contraception from screening through the last study visit: hormonal (oral, implant, or injection) begun >30 days prior to screening; barrier (condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD). Acceptable contraceptive options may also include abstinence, relationship with same sex partner or partner who has had a vasectomy at least six (6) months prior to the screening visit
3. Male subjects only: willing to use contraception or abstain from sexual activity beginning with the first exposure to study drug and continuing until discharged from the study due to completion or Early Termination
4. Healthy, as determined by the Investigator (in consultation with the Medical Monitor, as needed), based on medical and dental history, concurrent illnesses, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (extraoral, head and neck) during Screening Note: Subjects on a stable dose of medication may be eligible for screening and will be assessed by the Medical Monitor on a case-by-case basis.
5. Have a minimum of 12 bicuspids and molars with a minimum of 8 molars and bicuspids NOT having restorations, crowns, sealants
6. Demonstrated ability to expectorate ≥2 mL of stimulated saliva in 5 minutes
7. Have a salivary S. mutans of 1.0 x 10^5 colony forming units (CFUs)/mL or greater at Screening using mitis salivarius-bacitracin (MSB) agar plating
8. Willing to refrain from using non-study dentifrice and other non-study oral care products (oral care rinses, fluoride products, etc.) during the study
9. Willing to postpone elective dental procedures (e.g., dental cleanings) between Screening and final post-treatment visit (End of Study or Early Termination)
10. Willing and able to comply with oral hygiene and diet instructions
11. Has dentition adequate for custom dental tray gel application
12. Able to understand and sign the Assent and/or Informed Consent Form prior to initiation of study procedures
13. Able to communicate with the Investigator/study center personnel, understand and comply with the study requirements, and willing to return for protocol-specified visits at the appointed times

Exclusion Criteria:

1. Advanced periodontal disease
2. Active caries lesion(s) within 30 days prior to study drug administration (confirmed by comprehensive caries examination including standard radiographs if deemed necessary by the Investigator) Note: Subjects presenting with insipient, non-cavitated lesion(s) are not excluded
3. Medical condition (e.g., artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
4. Pathologic lesions of the oral cavity (suspicious or confirmed)
5. Full dentures or orthodontic appliances, e.g., braces; Note: partial dentures, removable retainers and night guards are not excluded, provided that they are cleaned regularly throughout the duration of the study.
6. Use of systemic antibiotics, topical oral antibiotics, or use of other drugs, which in the opinion of the Investigator could influence the study outcome, within 30 days prior to Screening and throughout the entire study.
7. Medical history indicating the woman is pregnant, breastfeeding/lactating or has a positive urine pregnancy test
8. Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to study drug administration (depending on the specifics, participation in an observational study is not necessarily excluded)
9. Prior participation in a C16G2 clinical trial and known to have received C16G2 active gel or mouth rinse Note: Placebo subjects are not excluded
10. Presence of any condition or concurrent illness, which in the opinion of the Investigator, would compromise normal immune function (e.g., diabetes, rheumatoid arthritis, lupus, liver disease, organ transplant, etc.), interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements, or jeopardize the safety of the subject or the validity of the study results

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Antimicrobial Activity of C16G2 | Evaluated over up to 5 months
  To assess the targeted antimicrobial activity of C16G2 Gel applications as measured by a reduction in Streptococcus mutans in saliva and dental plaque
Total Oral Bacterial Levels | Evaluated 7 days post last study drug administration
  Total bacterial levels will be evaluated by measuring cfu/ml counts of salivary and plaque bacteria
Safety of C16G2 Gel Administrations assessed by performing targeted physical examinations, oral cavity exams, taking vital signs and collection of adverse events | Up to 7 days post last study drug administration
  Safety will be assessed by performing targeted physical examinations, oral cavity exams, taking vital signs and collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wolff, DDS, PhD, Principal Investigator — NYU Langone Health
Locations (10):
- United States (10):
  - Imperial Beach Family Dentistry, Imperial Beach, California
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - Tufts University, Boston, Massachusetts
  - John F. Pittaway, DMD, Kalispell, Montana
  - Plaza West II Dental Group, Kalispell, Montana
  - New York University College of Dentistry, New York, New York
  - East Carolina University, Greenville, North Carolina
  - University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania
  - Texas Baylor College of Dentistry, Dallas, Texas
  - Anthony Henegar, DDS, PA, Irving, Texas